CLINICAL TRIAL: NCT04607382
Title: Patient Panel Survey on Menstrual Symptoms, HRQoL and Work Productivity in Patients With Primary or Secondary Dysmenorrhea in Japan
Brief Title: Survey on Menstrual Symptoms, Health Related Quality of Life and Work Productivity in Patients Suffering From Pain During Menstruation (Dysmenorrhea) in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21420
Record Dates: First submitted 2020-09-18; First posted 2020-10-29 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-dose estrogen progestin products (LEP): The patients in the LEP cohort should not have taken LEP in the last 2 months before the enrollment in the study, and will take LEP during the study period.
  Interventions: Drug: LEP
- Non-LEP: Those patients in the Non-LEP cohort should not have taken LEP in the last 2 months before the enrollment and will take NSAIDs and/or Chinese medicine (CM) during the study period.
  Interventions: Drug: NSAIDs and/or Chinese medicine (CM)

INTERVENTIONS:
Drug: LEP — LEP dosage up to the discretion of the treating gynecologists.
  Groups: Low-dose estrogen progestin products (LEP)
Drug: NSAIDs and/or Chinese medicine (CM) — Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) and Chinese medicine (CM) dosage up to the discretion of the treating gynecologists.
  Groups: Non-LEP

SUMMARY:
In this study researcher want to gain more information on the treatment effect of Low-dose Estrogen Progestin (a hormone treatment) on the health related quality of life and work productivity in patients suffering from menstrual pain. The treating doctors will ask the study participants to complete questionnaires at start of study, after 2 and 4 months (end of study). The questions will be about participant's general and mental health, concentration, behavioral and emotional changes, and work productivity and activity level. This study will be conducted in Japan and enrols about 380 female participants in the age range of 16 to 39 years.

ELIGIBILITY:
Female patients with a diagnosis of dysmenorrhea will be enrolled after the decision for treatment with LEP or Non-LEP has been made by the physician. Patients who have been prescribed LEP or Non-LEP for a medically appropriate use will be eligible to be enrolled. Indications and contraindications according to the local market authorization should be carefully considered. Evidence of assessment of all eligibility criteria by the patients, as well as enrollment of a patient in the study should be documented in database of M3.

Inclusion Criteria:

Patients who meet all the inclusion criteria will be enrolled in this study.

* Patients between the ages of 16 and 39
* Patients diagnosed with primary or secondary dysmenorrhea by gynecologists
* Patients who can visit ob/gyn clinics or hospitals every 6 months to have consultations with gynecologists for treatment of dysmenorrhea
* Patients who plan to be treated with drug for dysmenorrhea after enrollment in this study
* Patients who are currently on Non-LEP therapies will be eligible for LEP cohort**
* Patients who can access the website to complete the questionnaire using mobile communication equipment such as mobile phones or tablets
* Patients who submit an informed consent on the website before the start of this study

Exclusion Criteria:

Patients who meet any of the exclusion criteria will not be enrolled in this study.

* Patients who have taken LEP for dysmenorrhea in the last 2 months before enrollment*
* Patients with mental disorders such as depression, severe infectious diseases, or malignant tumors
* Patients who do not meet the inclusion criteria.

Patients with contraindications for LEP or COC are as follows:

* Women who have a predisposition to hypersensitivity to the ingredients of this product
* Breast cancer patients
* Patients with undiagnosed abnormal genital bleeding
* Patients with thrombophlebitis, pulmonary embolism, cerebrovascular disease, coronary artery disease, or a history of the same
* Smokers over the age of 35 who smoke more than 15 cigarettes a day
* Patients with migraine with antecedents (flashing lights, star-shaped flashes, etc.)
* Patients with valvular heart disease complicated by pulmonary hypertension or atrial fibrillation and with a history of subacute bacterial endocarditis
* Diabetic patients with vascular lesions (diabetic nephropathy, diabetic retinopathy, etc.)
* Patients with thrombotic predisposition
* Patients with antiphospholipid antibody syndrome
* Patients with major surgeries of 30 minutes or more, within 4 weeks before surgery, within 2 weeks after surgery, and in patients with long-term rest
* Patients with severe liver damage.
* Patients with liver tumors
* Hypertension (except for patients with mild hypertension)
* Otosclerosis
* Patients with a history of jaundice, persistent pruritus, or herpes pregnancy during pregnancy
* Women who are pregnant or who may be pregnant
* Breastfeeding women under 6 months of age
* Patients taking contraindicated drugs for LEP or COC

Ages: 16 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The study is a prospective, non-interventional study for patients being treated for primary or secondary dysmenorrhea in real-world clinical practice. Patients will be recruited using M3 group network. M3 is a company that provides a medical portal site for HCPs, and more than 280,000 medical doctors are registered with M3 with 80% coverage in Japan. As many patients with dysmenorrhea visit ob/gyn clinics rather than hospitals, patients diagnosed as primary or secondary dysmenorrhea will be recruited by gynecologists who work in the clinics enrolled in M3. When patients agree to participate in the study, the gynecologists provide the QR code or URL to the patients enabling them to access the site from their mobile communication equipment such as mobile phones and tablets, and answer the questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Menstrual Distress: evaluated by modified Menstrual Distress Questionnaire (mMDQ) | Baseline, 60 days and 120 days
  To describe the changes in menstrual symptoms before, during and after the study in Low-dose Estrogen Progestin product (LEP) cohort.
Changes in Health Related Quality of Life (HRQoL): evaluated by Short Form (36) Health Survey version 2 (SF-36v2) | Baseline, 60 days and 120 days
  To describe the changes in HRQoL before, during and after the study in LEP cohort.
  The SF-36v2 will be assessed on a 3- and 5-point Likert scale. The rating scale depends on each question.
Changes in work productivity (mWPAI) | Baseline, 60 days and 120 days
  To describe the changes in work productivity before, during and after the study in LEP cohort.
Changes in Activity Impairment: evaluated by General Health v2.0 (WPAI-GH) | Baseline, 60 days and 120 days
  To describe the changes in activity impairment before, during and after the study in LEP cohort.

SECONDARY OUTCOMES:
Description of patients' background and medical history of LEP and Non-LEP cohorts | Baseline
  To describe patients' background and medical history of LEP and Non-LEP cohorts
Change in mMDQ of Non-LEP cohort | Baseline, 60 days and 120 days
  To describe the change in menstrual symptoms before, during and after the study in Non-LEP cohort.
Change in HRQoL of Non-LEP cohort | Baseline, 60 days and 120 days
  To describe the change in HRQoL before, during and after the study in Non-LEP cohort.
Change in work productivity of Non-LEP cohort | Baseline, 60 days and 120 days
  To describe the change in work productivity before, during and after the study in Non-LEP cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Facilities, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Yoshino O, Takahashi N, Suzukamo Y. Menstrual Symptoms, Health-Related Quality of Life, and Work Productivity in Japanese Women with Dysmenorrhea Receiving Different Treatments: Prospective Observational Study. Adv Ther. 2022 Jun;39(6):2562-2577. doi: 10.1007/s12325-022-02118-0. Epub 2022 Apr 1. PMID 35362862